CLINICAL TRIAL: NCT07314372
Title: A Prospective Phase II Study of Fatty Acid Degradation (FAD) Subtype-Guided Comprehensive Therapy for Unresectable Hepatocellular Carcinoma
Brief Title: FAD Subtype-Guided Combination Therapy for Unresectable Hepatocellular Carcinoma
Acronym: FAD-HCC-001
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, YU DE CAI, Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAD-HCC-001
Record Dates: First submitted 2025-11-22; First posted 2026-01-02 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Unresectable Hepatocellular Carcinoma (HCC); Hepatocellular Carcinoma (HCC); Liver Cancer Adult
Keywords: Hepatocellular Carcinoma; Fatty Acid Degradation; Metabolic Subtyping; Precision Medicine; Conversion Therapy; Immunotherapy; Anti-angiogenic Therapy; TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- F1/F2 Subtype: Camrelizumab Plus Apatinib (Experimental): Participants whose tumors are classified as F1 or F2 based on the fatty acid degradation (FAD) subtype will receive systemic therapy with camrelizumab and apatinib. Camrelizumab is administered intravenously at 200 mg every 3 weeks, and apatinib is taken orally at 250 mg once daily. Treatment continues until disease progression, unacceptable toxicity, withdrawal of consent, or completion of the planned treatment duration. Imaging assessments are conducted every 6 weeks to evaluate tumor response.
  Interventions: Drug: Camrelizumab Plus Apatinib
- F3 Subtype: TACE Plus Camrelizumab and Apatinib (Experimental): Participants with the F3 metabolic subtype, characterized by high fatty acid degradation activity, will receive transarterial chemoembolization (TACE) in addition to systemic therapy. Camrelizumab (200 mg IV every 3 weeks) and apatinib (250 mg orally once daily) are administered on the same schedule as the F1/F2 arm. TACE is performed 2-4 weeks after systemic therapy initiation, with up to two treatments per tumor (maximum four sessions total). Apatinib is paused 3-5 days before TACE and restarted 3-5 days afterward. Treatment continues until disease progression, unacceptable toxicity, or discontinuation for clinical reasons. Imaging assessments occur every 6 weeks.
  Interventions: Drug: TACE Plus Camrelizumab and Apatinib

INTERVENTIONS:
Drug: Camrelizumab Plus Apatinib — Camrelizumab is administered intravenously at 200 mg every 3 weeks, and apatinib is taken orally at 250 mg once daily.
  Arms: F1/F2 Subtype: Camrelizumab Plus Apatinib
Drug: TACE Plus Camrelizumab and Apatinib — Camrelizumab (200 mg IV every 3 weeks) and apatinib (250 mg orally once daily) are administered on the same schedule as the F1/F2 arm. TACE is performed 2-4 weeks after systemic therapy initiation, with up to two treatments per tumor (maximum four sessions total). Apatinib is paused 3-5 days before TACE and restarted 3-5 days afterward.
  Arms: F3 Subtype: TACE Plus Camrelizumab and Apatinib

SUMMARY:
This study is a prospective, multicenter Phase II trial evaluating a personalized treatment strategy for patients with unresectable hepatocellular carcinoma (HCC). The study uses a metabolic classification system called the fatty acid degradation (FAD) subtype to guide therapy selection. Patients will be assigned to different treatment groups based on their tumor's FAD subtype, determined through RNA-seq analysis of the tumor tissue obtained from liver biopsy.

DETAILED DESCRIPTION:
This prospective, multicenter Phase II study evaluates a precision-medicine treatment strategy for unresectable hepatocellular carcinoma (HCC) using a metabolic classification system based on fatty acid degradation (FAD). Prior translational research has shown that HCC exhibits heterogeneous metabolic phenotypes, and that tumors with distinct FAD signatures demonstrate different immune microenvironments and therapeutic sensitivities. Building on these findings, this study applies FAD subtype profiling in clinical practice to guide individualized treatment selection.

All enrolled patients will undergo tumor tissue analysis for transcriptomic assessment and FAD scoring. When tumor tissue is not immediately obtainable, MRI fat-fraction measurement may be used temporarily to facilitate enrollment, with tissue-based classification performed afterward. Based on the predefined FAD subtypes (F1, F2, and F3), patients will be allocated to tailored therapeutic strategies designed to align with each subtype's metabolic and microenvironmental characteristics.

Patients with F1 or F2 subtypes will receive systemic therapy with camrelizumab and apatinib, reflecting prior evidence that these subtypes may benefit from immunotherapy combined with anti-angiogenic therapy. Patients with the F3 subtype that characterized by enhanced lipid metabolic activity will receive TACE in addition to camrelizumab and apatinib.

Treatment is delivered in 3-week cycles, with imaging assessments performed regularly to evaluate tumor response. Safety will be closely monitored throughout the study, including immunotherapy-related toxicities, anti-angiogenic drug-associated events, and TACE-related complications. After discontinuation of study treatment, participants will enter a structured follow-up schedule to monitor survival and subsequent treatments.

In addition to evaluating clinical outcomes, the study incorporates exploratory biomarker analyses, including transcriptomics, metabolomics, and imaging-based fat quantification. These analyses aim to improve understanding of how metabolic subtypes influence therapeutic response and resistance mechanisms, and to assess whether MRI-based fat fraction can serve as a noninvasive surrogate for molecular FAD classification.

Overall, this study seeks to translate metabolic phenotyping into clinical decision-making and to determine whether FAD-guided personalized therapy can improve treatment outcomes for patients with unresectable HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age who voluntarily agree to participate and sign informed consent.
2. Histologically or cytologically confirmed hepatocellular carcinoma (HCC).
3. Unresectable or not suitable for curative local therapy, or progression after prior surgery or local therapy.
4. BCLC stage B or C.
5. No prior systemic therapy for HCC.
6. At least one measurable lesion according to RECIST v1.1.
7. Availability of fresh or archival tumor tissue for FAD subtype testing; if not available at screening, MRI fat fraction may be used temporarily.
8. Child-Pugh class A or B (≤7 points).
9. ECOG performance status 0-1.
10. Adequate organ function, including:

    * ANC ≥1.5 × 10⁹/L
    * Platelets ≥75 × 10⁹/L
    * Hemoglobin ≥90 g/L
    * Albumin ≥30 g/L
    * Total bilirubin ≤1.5 × ULN
    * ALT and AST ≤3 × ULN
    * Serum creatinine ≤1.5 × ULN or creatinine clearance >50 mL/min
    * INR ≤1.2 or PT within 2 seconds above ULN
    * Urine protein <2+ or 24-hour urine protein <1.0 g
11. Controlled HBV infection (HBV-DNA <2000 IU/mL; if above this level, ≥1 week of antiviral therapy with ≥1-log reduction prior to first dose). HCV-positive individuals must be managed per clinical guidelines.
12. Life expectancy ≥12 weeks.
13. Women of childbearing potential must have a negative pregnancy test; participants of reproductive potential must agree to effective contraception during treatment and for 6 months afterward.

Exclusion Criteria:

1. Non-HCC primary liver cancers (e.g., cholangiocarcinoma, combined HCC-CCA).
2. F3 subtype without liver lesions on imaging.
3. Clinically significant ascites requiring therapeutic intervention, or uncontrolled pleural/pericardial effusion.
4. Interstitial lung disease, pneumonitis requiring steroids, or active pulmonary infection.
5. Active or history of autoimmune disease requiring systemic treatment (exceptions allowed per protocol, e.g., controlled hypothyroidism).
6. Recent use (within 2 weeks) of systemic immunosuppressive therapy >10 mg/day prednisone equivalent.
7. Gastrointestinal bleeding within 6 months, high-risk varices, active ulcers, fistula, perforation, or intra-abdominal abscess.
8. Known bleeding or clotting disorders; therapeutic anticoagulation not permitted.
9. Thromboembolic events within 6 months (e.g., stroke, PE).
10. Significant cardiovascular disease, including NYHA class ≥II heart failure, recent MI (within 1 year), unstable angina, clinically significant arrhythmias, or QTc prolongation.
11. Uncontrolled hypertension (SBP ≥140 mmHg or DBP ≥90 mmHg despite treatment), or history of hypertensive crisis.
12. Major vascular disease within 6 months (e.g., arterial thrombosis, aneurysm requiring repair).
13. Serious non-healing wounds, active ulcers, or fractures.
14. Inability to swallow oral medication or conditions affecting drug absorption.
15. Severe infection within 4 weeks, therapeutic antibiotics within 14 days, fever ≥38.5°C within 7 days before enrollment, or WBC >15 × 10⁹/L.
16. Known HIV infection or other causes of immunodeficiency.
17. Receipt of live attenuated vaccines within 28 days before treatment.
18. Any condition that, in the investigator's judgment, would interfere with study participation or interpretation of results, including substance abuse, severe psychiatric illness, or social factors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From first dose until first documented disease progression or death, whichever occurs first, assessed up to 24 months.
  ORR is defined as the proportion of participants who achieve a confirmed complete response (CR) or partial response (PR) according to RECIST v1.1, as assessed by imaging every 6 weeks. ORR will be calculated separately for each FAD subtype cohort (F1/F2 and F3).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) by mRECIST | From first dose until first documented disease progression or death, whichever occurs first, assessed up to 24 months.
  ORR defined as the proportion of participants achieving complete response or partial response according to mRECIST criteria.
Disease Control Rate (DCR) | From first dose until first documented disease progression or death, whichever occurs first, assessed up to 24 months.
  DCR is defined as the proportion of participants achieving complete response, partial response, or stable disease according to RECIST v1.1.
Progression-Free Survival (PFS) | From first dose until radiographic disease progression or death, whichever occurs first, assessed up to 24 months.
  PFS will be estimated using RECIST v1.1 criteria and assessed every 6 weeks.
Overall Survival (OS) | From first dose until death from any cause, assessed up to 24 months.
  OS is defined as the time from study treatment initiation to death from any cause.
Duration of Response (DoR) | From first documented response (CR or PR) until disease progression or death, whichever occurs first, assessed up to 24 months.
  DoR applies to participants achieving CR or PR per RECIST v1.1.
Conversion-to-Surgery or Local Ablative Therapy Rate | Throughout study treatment, up to 24 months
  Proportion of participants converted from unresectable to resectable disease or eligible for curative local therapy based on multidisciplinary assessment.
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From first dose through 90 days after last dose
  Safety will be evaluated according to CTCAE v5.0; TACE-related complications will be described separately for the F3 cohort.

OTHER OUTCOMES:
Correlation Between MRI-Derived Fat Fraction and Transcriptomic FAD Subtype Score | From baseline tissue/MRI assessment until end of treatment, assessed up to 24 months.
  This outcome measure evaluates the correlation between tumor fat content measured by MRI and fatty acid degradation (FAD) activity determined by transcriptomic analysis. MRI fat fraction (FF): Quantified as percentage (%) of intra-tumoral fat content, measured using chemical shift-encoded MRI.
  FAD subtype score: Quantified as a continuous FAD score calculated from RNA sequencing-based transcriptomic data using single-sample gene set enrichment analysis (ssGSEA).
  Correlation analysis will be performed between MRI-derived fat fraction percentage and the transcriptomic FAD score to assess the concordance between imaging-based and molecular-based FAD classification.
Correlation Between Molecular Biomarker Levels and Objective Tumor Response | Baseline, on-treatment, and at disease progression (up to 24 months)
  This outcome measure evaluates the correlation between molecular biomarker levels and objective tumor response.
  Transcriptomic biomarkers: Gene expression levels measured in tumor tissue by RNA sequencing (RNA-seq) and expressed as normalized gene expression values.
  Metabolomic biomarkers: Relative metabolite levels measured in blood or tumor tissue by mass spectrometry-based metabolomic profiling, expressed as relative abundance units.
  Objective tumor response: Measured by RECIST v1.1 using CT or MRI and expressed as response status (complete response or partial response vs. no response).
  Correlation analyses will be performed between each molecular biomarker measurement (gene expression values, metabolite abundance) and objective tumor response.
Correlation Between Molecular Biomarker Levels and Treatment Response | From baseline until disease progression, assessed up to 24 months.
  This measure evaluates the correlation between molecular biomarker levels and treatment response. Biomarker levels will be quantified using:
  Transcriptomic profiling: Gene expression levels measured by RNA sequencing (RNA-seq) and expressed as normalized expression counts.
  Metabolomic profiling: Relative metabolite concentrations measured by untargeted mass spectrometry, expressed as relative abundance units.
  Treatment response will be defined using RECIST v1.1. Correlation analyses will be conducted between each biomarker measurement (gene expression counts and metabolite abundance) and tumor response outcomes.
Correlation Between FAD Metabolic Subtype and Clinical Outcomes | Up to 36 months
  This outcome measure evaluates the correlation between the fatty acid degradation (FAD) metabolic subtype and overall survival (OS) or progression-free survival (PFS).
  FAD metabolic subtype: Classified as F1, F2, or F3 using RNA sequencing-based transcriptomic analysis with ssGSEA scoring.
  Overall Survival (OS): Measured in months, defined as the time from initiation of study treatment until death from any cause.
  Progression-Free Survival (PFS): Measured in months, defined as the time from initiation of study treatment to radiographic disease progression or death, assessed by RECIST v1.1 using CT or MRI imaging.
  Correlation analyses will be performed between FAD subtype classification and OS/PFS duration.

CONTACTS AND LOCATIONS:
Overall Officials: Decai Yu, Doctor, Study Chair — the Affiliated Drum Tower Hospital, Medical School of Nanjing University
Locations (1):
- Nanjing Drum Tower Hospital, The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The study involves genomic, transcriptomic, and clinical imaging data that may pose risks to participant privacy, and data sharing is not planned.

REFERENCES:
- [Background] Li B, Wen J, Xu Z, Yan P, Han B, Yu D. Comprehensive analysis of transcriptomic biomarkers for predicting response to atezolizumab plus bevacizumab immunotherapy in hepatocellular carcinoma. Clin Mol Hepatol. 2025 Jan;31(1):e31-e34. doi: 10.3350/cmh.2024.0628. Epub 2024 Sep 20. No abstract available. PMID 39300923
- [Background] Li B, Li Y, Zhou H, Xu Y, Cao Y, Cheng C, Peng J, Li H, Zhang L, Su K, Xu Z, Hu Y, Lu J, Lu Y, Qian L, Wang Y, Zhang Y, Liu Q, Xie Y, Guo S, Mehal WZ, Yu D. Multiomics identifies metabolic subtypes based on fatty acid degradation allocating personalized treatment in hepatocellular carcinoma. Hepatology. 2024 Feb 1;79(2):289-306. doi: 10.1097/HEP.0000000000000553. Epub 2023 Aug 7. PMID 37540187